CLINICAL TRIAL: NCT05145868
Title: Evaluation and Optimization of a Just-in-Time Messaging Intervention to Reduce Alcohol-Facilitated Intimate Partner Violence Perpetration Among At-Risk Young Adult Men and Women
Brief Title: Just-In-Time Intervention to Reduce Alcohol-Facilitated Intimate Partner Violence Perpetration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Cynthia Stappenbeck, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP00014947
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Drinking; Aggression; Emotion Regulation
MeSH Terms: conditions — Alcohol Drinking; Aggression; Emotional Regulation | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive the RELATE intervention.
  Interventions: Behavioral: Alcohol Skills and Emotion Regulation Intervention
- Attention Control (Active Comparator): Participants in this arm will receive supportive control messages.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Alcohol Skills and Emotion Regulation Intervention — The text-based intervention will provide alcohol reduction strategies and emotion regulation skills.
  Arms: Intervention
Other: Attention Control — Text-messages will be sent that include no intervention content to serve as an attention control
  Arms: Attention Control

SUMMARY:
Acute alcohol intoxication is a robust predictor of intimate partner violence (IPV) perpetration for young adult men and women; therefore, interventions delivered proximally to drinking episodes - a period of high risk - are needed to reduce alcohol-facilitated IPV. This project seeks to improve public health by delivering a just-in-time text messaging intervention proximally to drinking episodes and evaluating the impact of the intervention on alcohol-facilitated IPV in a sample of at-risk young adult men and women. Additionally, through an innovative design this project is poised to answer these important questions: whether receiving a message, when, for whom, what type, and under what conditions this just-in-time messaging intervention leads to reductions in alcohol use and IPV perpetration.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* Consumed alcohol an average of 2 times per week in last 3 months
* At least two instances of heavy episodic drinking in last month
* Currently in a romantic relationship
* History of IPV perpetration within last 3 months
* Willing to provide cell phone number and carrier and receive text messages for 30 days

Exclusion Criteria:

* None

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use | 30 days
  Drinking Quantity (number of drinks consumed)
Alcohol Use | 1-month follow-up
  Drinking Quantity (number of drinks consumed)
Alcohol Use | 3-month follow-up
  Drinking Quantity (number of drinks consumed)
Alcohol Use | 6-month follow-up
  Drinking Quantity (number of drinks consumed)
Intimate Partner Violence | 30 days
  Occurrence (yes/no) of psychological or physical Aggression against an intimate partner
Intimate Partner Violence | 1-month follow-up
  Frequency of Psychological or Physical Aggression against an intimate partner
Intimate Partner Violence | 3-month follow-up
  Frequency of Psychological or Physical Aggression against an intimate partner
Intimate Partner Violence | 6-month follow-up
  Frequency of Psychological or Physical Aggression against an intimate partner

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stappenbeck, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States